CLINICAL TRIAL: NCT00123435
Title: Does Step Count Feedback Enhance Counseling for Weight Loss?
Brief Title: Veterans Walk for Health Study
Acronym: VWH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D3358-R
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Hyperlipidemia; Hypertension; Obesity
Keywords: Behavioral Research; Nutritional management; Physical activity; Prevention; Randomized control trial; walking program; Weight loss; World wide web
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hyperlipidemias; Hypertension; Obesity; Motor Activity; Weight Loss | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): 5-session nutritional counseling program
  Interventions: Behavioral: Nutritional counseling; Behavioral: Walking program
- Arm 2 (Experimental): 5-session nutritional counseling program + simple pedometer feedback
  Interventions: Behavioral: Nutritional counseling; Behavioral: Walking program; Device: Simple pedometer
- Arm 3 (Experimental): 5-session nutritional counseling program + simple pedometer feedback + enhanced pedometer feedback web-based feedback
  Interventions: Behavioral: Nutritional counseling; Behavioral: Walking program; Device: Simple pedometer; Device: Enhanced pedometer

INTERVENTIONS:
Behavioral: Nutritional counseling — The nutritional counseling is based on the six-session Medical Nutrition Therapy Protocol for Weight Management published by the American Dietetics Association. The categories include the following: a) Meal planning (food, hydration, fiber, alcohol), b) Food label reading, c) Recipe modification, d) Food preparation, e) Dining out and f) Physical activity.
  Arms: Arm 1
Behavioral: Walking program — As part of the discussion of physical activity, participants in the control group will be encouraged to walk and dietitians will discuss goal setting using timed walks instead of total daily step-counts at each of the control group sessions. As a general guideline, participants will be encouraged to increase their daily walking target by 5-10 minutes (control group with time goals) or to increase their average daily step counts by 10-25% (pedometer group with step count goals) following each of the nutritional counseling sessions.
  Arms: Arm 1
Behavioral: Nutritional counseling — The nutritional counseling is based on the six-session Medical Nutrition Therapy Protocol for Weight Management published by the American Dietetics Association. The categories include the following: a) Meal planning (food, hydration, fiber, alcohol), b) Food label reading, c) Recipe modification, d) Food preparation, e) Dining out and f) Physical activity.
  Arms: Arm 2
Behavioral: Walking program — As part of the discussion of physical activity, participants in the control group will be encouraged to walk and dietitians will discuss goal setting using timed walks instead of total daily step-counts at each of the control group sessions. As a general guideline, participants will be encouraged to increase their daily walking target by 5-10 minutes (control group with time goals) or to increase their average daily step counts by 10-25% (pedometer group with step count goals) following each of the nutritional counseling sessions.
  Arms: Arm 2
Device: Simple pedometer — Device to be worn during waking hours to give an objective measure of steps taken each day.
  Arms: Arm 2
Behavioral: Nutritional counseling — The nutritional counseling is based on the six-session Medical Nutrition Therapy Protocol for Weight Management published by the American Dietetics Association. The categories include the following: a) Meal planning (food, hydration, fiber, alcohol), b) Food label reading, c) Recipe modification, d) Food preparation, e) Dining out and f) Physical activity.
  Arms: Arm 3
Behavioral: Walking program — As part of the discussion of physical activity, participants in the control group will be encouraged to walk and dietitians will discuss goal setting using timed walks instead of total daily step-counts at each of the control group sessions. As a general guideline, participants will be encouraged to increase their daily walking target by 5-10 minutes (control group with time goals) or to increase their average daily step counts by 10-25% (pedometer group with step count goals) following each of the nutritional counseling sessions.
  Arms: Arm 3
Device: Simple pedometer — Device to be worn during waking hours to give an objective measure of steps taken each day.
  Arms: Arm 3
Device: Enhanced pedometer — Simple pedometer with the addition of web-based feedback.
  Arms: Arm 3

SUMMARY:
The objective of this study is to determine whether a tailored web-based system for providing feedback on walking step-counts, in combination with regular nutrition counseling, can improve weight loss over nutrition counseling alone in patients with heart disease.

DETAILED DESCRIPTION:
Objective: This proposal was developed at the request of, and with input from, the Research Council of the Department of Veterans Affairs' (VA's) National Advisory Board for Nutrition and Food Services, in an effort to address obesity, a major health problem for VA patients. The prevalence of obesity in the United States has been increasing at an alarming rate. As a result, obesity related chronic diseases such as diabetes are also increasing in prevalence. While interventions that focus only on dietary changes can result in significant weight loss, the lost weight is often rapidly regained. Physical activity, when added to a dietary weight loss program, not only increases the initial weight loss but it also can play a critical role in preventing weight regain. The primary objective of the proposed study is to test the efficacy of a low-cost, innovative weight loss program targeting lifestyle physical activity and diet in individuals with cardiovascular risk factors or disease.

Study Design and Methods: In this 3 year multi-site randomized controlled trial, the investigators will recruit overweight and obese veterans with cardiovascular disease risk factors or known cardiovascular disease who have been referred for nutritional counseling or who have responded to advertisements for the study. Research participants will be randomized to one of three study groups:

* nutritional counseling alone;
* nutritional counseling with simple pedometer feedback; and
* nutritional counseling, with both simple pedometer and enhanced pedometer (web-based) feedback.

Each participant will have 5 visits with a dietitian in the course of 6 months. Participants randomized to receive pedometer feedback will review objectively monitored step-count data during their nutritional counseling sessions and will use the data to set new step-count goals. The primary outcome, weight loss, will be assessed at the sixth and final session at the end of the 6-month intervention. Enhanced pedometers that can monitor step-counts throughout the day and upload time stamped step count data to a central computer will be used to monitor adherence to a walking program.

ELIGIBILITY:
Inclusion Criteria:

* Is newly referred from a VA physician for nutritional counseling or has responded to an advertisement for the study - Has one of the following diagnoses: diabetes, coronary artery disease, hypercholesterolemia, hypertension, obesity.
* Is ambulatory and able to comfortably walk at least one block.
* Has a body mass index (BMI) of 28 or greater.
* Is not already regularly active (30 minutes a day, 5 days a week of moderate intensity physical activity).
* Is in the contemplation or preparation stage of readiness to become more physically active.
* Is willing to try a walking program.
* Can communicate comfortably in English.

Exclusion Criteria:

* Has attended a nutritional counseling session in the past 28 days.
* May be at risk for adverse cardiovascular events with a walking program--specifically participants who:

  * have symptoms of cardiovascular disease (CVD) while walking;
  * have been told by a physician that walking might be dangerous; or
  * have a stress test scheduled in the next two months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2005-07; Primary Completion 2007-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | week 2, week 3, week 6, week 12, and week 24

SECONDARY OUTCOMES:
Average daily activity level | week 2, week 12, and week24
Quality of life and participant satisfaction | week 1, week 12, and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Richardson, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Julie C Lowery, PhD MHSA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Goodrich DE, Larkin AR, Lowery JC, Holleman RG, Richardson CR. Adverse events among high-risk participants in a home-based walking study: a descriptive study. Int J Behav Nutr Phys Act. 2007 May 23;4:20. doi: 10.1186/1479-5868-4-20. PMID 17521443